CLINICAL TRIAL: NCT05596058
Title: Efficacy of a Non-pharmacological Treatments on Neurophysiological and Clinical Outcomes
Brief Title: Non-pharmacological Treatments in Migraine.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the unavailability of the subjects who gave the consent to participate to the study protocol
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Manuela Deodato, Principal Investigator, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080_2020
Record Dates: First submitted 2022-05-23; First posted 2022-10-27 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Migraine
Keywords: Migraine; Habituation; Sensitization; transcranial Magnetic stimulation
MeSH Terms: conditions — Migraine Disorders; Substance-Related Disorders | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: We are going to use a simple randomization scheme 1:1:1 with excel and assign subjects into three groups respectively: 15 patients in physical-cognitive tasks groups, 15 patients in active exercise Only and 15 patients in Cognitive training.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients do not know other type of intervention; who have to do the assessment do not know the type of interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual task (active exercise and cognitive task) (Experimental): The dual task protocol is going to be in 15 one-hour sessions once a week in the headache free days.
  This protocol will be set up in the clinic of physiotherapy degree (University of Trieste in the Department of Medical, Surgical, and Health Sciences).
  The physical training tasks will be associated with concomitant cognitive tasks specifically relying on executive function.
  The goal is to engage the three core executive functions: inhibition (the ability to inhibit automated responses), working memory (the ability to hold, process, and manipulate information in mind) and shifting (the ability to change stimulus-response associations for performing an ongoing task).
  Patients will be exposed to different cognitive tasks during physical activity such as walking or running on the treadmill, indoor cycling and balance exercises.
  -
  Interventions: Other: dual task protocol: active exercises with concomitant cognitive training in executive functions
- active exercise only (Active Comparator): The active exercise only intervention is going to consist of aerobic and flexibility training with a targeted duration of 1 hour, twice per week for 3 months.
  Interventions: Other: active exercise
- Cognitive task trainig only (Active Comparator): The Cognitive task training only engage the three core executive functions: inhibition (the ability to inhibit automated responses), working memory (the ability to hold, process, and manipulate information in mind) and shifting (the ability to change stimulus-response associations for performing an ongoing task).
  Interventions: Other: cognitive task only

INTERVENTIONS:
Other: dual task protocol: active exercises with concomitant cognitive training in executive functions — The active exercise tasks will be associated with concomitant cognitive tasks specifically relying on executive function.
  The goal is to engage the three core executive functions: inhibition (the ability to inhibit automated responses), working memory (the ability to hold, process, and manipulate information in mind) and shifting (the ability to change stimulus-response associations for performing an ongoing task).
  Patients will be exposed to different cognitive tasks during physical activity such as walking or running on the treadmill, indoor cycling and balance exercises.
  Arms: Dual task (active exercise and cognitive task)
Other: active exercise — Physical activity and motor task only
  Arms: active exercise only
Other: cognitive task only — cognitive exercise in executive functions
  Arms: Cognitive task trainig only

SUMMARY:
Migraine may have an adverse effect on physical, cognitive, and psychosocial functioning. It causes major consequences for the quality of life of the sufferer and a major burden on the health care system.

About the physiopathology, two opposing processes, depression (habituation) and facilitation (sensitization), determine the final behavioural outcome after a sequence of repetitive stimuli.

Sensitization is a general behavioural response of augmentation to innocuous sensory and noxious stimuli. It has been associated with a dysfunction in descending pain inhibition.

The nature or intensity of a painful event does not strongly relate to the development of chronic pain, but an individual's behavioural response to the event contributes to chronicity. Imaging data have identified that chronic pain may change the structure of the brain in response to environmental demands.

It suggests that the brain of healthy control has a "healthy response" to frequent nociceptive input, such as "habituation", while chronic pain patients show a "maladaptive plasticity".

Habituation is "a response decrement as a result of repeated stimulation". It is a phenomenon observed in the autonomic and behavioural component called the "orienting response" in humans. The orienting response is elicited when a novel stimulus is encountered, and it directs attention toward that stimulus. When the same stimulus is presented repeatedly occur habituation. Researchers have found a number of physiological mechanisms associated with Orienting response. Habituation of the orienting response is a simple form of learning and acts an attentional filtering mechanism that makes people able to select what is part of their present goal and adapt to environment. In this way only one channel of information to be processed, with the rest filtered out. Habituation depends on a memory process whereby the organism learns to associate goal irrelevant stimuli with a no-consequence response.

Lack of Habituation during stimulus repetition is a functional property of the brain in people with migraine between attacks. Thalamo-cortical dysrhythmia and lack of H characterize migraineurs' brains. This abnormal information processing increases during the pain-free days, the vertex is just before the attack, and decreases in the ictal phase. Migraineurs are characterized by a generally increased sensitivity to visual (sensitivity to light), auditory (to sound), or somatic stimuli not only during the attack, but also outside of the attack.

It was confirmed also by analysing motor cortex excitability. Aerobic exercises may be effective as pharmacological treatment in the management of migraine and focused attention task may help human subjects to better ignore irrelevant stimuli.

The main aim of this study is to assess the efficacy of a non-pharmacological treatment, such as physical therapy, with a specific dual task protocol of active exercise with concomitant cognitive tasks, in relation to habituation (Transcranial magnetic stimulation) and sensitization (Algometer assessment) neurophysiological outcomes. The second aim is to assess these non-pharmacological treatments concerning to clinical outcomes (intensity of pain, duration of attacks and frequency of pain; neurophysiological test on executive functions).

DETAILED DESCRIPTION:
A Randomized Controlled Trial (RCT) will be conducted on three groups of patients with migraine. The project was approved by the institutional review board C.E.U.R. . Patients will be recruited and randomized by the Neurologic Clinic, Headache Centre (University of Trieste in the Department of Medical, Surgical, and Health Sciences), diagnosing Migraine after a neurologic visit (diagnostic criteria of ICDH3-beta).

In the first enrollment visit (T0), the patients will be undergone anamnestic evaluation, neurological and general objective examination. The following criteria of exclusion are going to be respected: pregnancy; serious psychiatric pathologies, serious pathologies as traumas, cancers or infective pathologies, important surgery procedures during the last year; physiotherapy and other no pharmacological treatment for another pathology; less than 18 years of age; presence of multiple migraine; presence of therapeutics changes linked to headache in the last 3 months; absence of pharmacological prophylaxis treatment in the last 3 months; no auditory or visual processing disorders. While, the criteria of inclusion are going to be the following: diagnosis migraine (diagnostic criteria of ICDH3-beta); Age over 18. Patients are going to be given a diary for cephalic outcome: frequency (headache days a month), intensity and duration of attack. The paper diary is going to inserted into a specific database for subsequent data analysis.

All patients are going to re-evaluated with the diary after one month (T1). The frequency is going to be between 15 days a month and 18 days a month. Transcranial magnetic Stimulation is going to be recorded.The Migraine disability assessment scale (MIDAS) will be performed. The MIDAS questionnaire consist of five questions aimed at assessing the impact of migraine on the patients' daily life in the 3 months prior to the study, in terms of absence from work or school, inability to carry out household chores, or take part in family, social, or leisure activities expressed in days. The final score was obtained by adding up the total number of days for each of the five questions.

Simple randomization scheme 1:1:1 was used with excel and assign subjects into three groups respectively: 15 patients in physical-cognitive tasks groups, 15 patients in active exercise Only and 15 patients in Cognitive task only. All patient going to sign the informed consent.

Patients will be allowed to take symptomatic medications in case of severe headache according to guidelines of the International Headache Society. Patients will be only asked to limit symptomatic medications consumption for a maximum twice per week in order to not affect the interpretation of data. Finally, after three months of treatment, the final visit will be performed (T2) with clinical re-evaluation of the patients and analysis of the cephalic parameters reported in the diary, the data of transcranial magnetic stimulation and the headache-related disability with MIDAS.

All patients will be reexamined at 1 months follow up (T3) with the diary, Transcranial magnetic stimulation and MIDAS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis migraine (diagnostic criteria of ICDH3-beta)
* Age over 18

Exclusion Criteria:

* pregnancy
* serious psychiatric pathologies
* serious pathologies as traumas, cancers or infective pathologies
* important surgery procedures during the last year
* physiotherapy and other no pharmacological treatment for another pathology
* less than 18 years of age;
* presence of multiple migraine
* presence of therapeutics changes linked to headache in the last 3 months
* absence of pharmacological prophylaxis treatment in the last 3 months
* no auditory or visual processing disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Values of Transcranial magnetic stimulation in migraine patients | Before each treatment
  Rest motor threshold in mV
Change from Baseline of the values of Transcranial magnetic stimulation in migraine patients at 3 months | 3 months
  Rest motor threshold in mV
Change from baseline of the value of Transcranial magnetic stimulation in migraine patients at 4 months | 4 months
  Rest motor threshold mV

SECONDARY OUTCOMES:
Headache parameters and MIDAS | Before each treatment
  migraine days per month assessed with diary
Headache parameters and MIDAS | 3 months of each treatment
  Change from baseline of migraine days per month assessed with diary at 3 months
Headache parameters and MIDAS | 4 months
  Change migraine days per month assessed with diary at 4 months
Algometer Assessment | Before each treatment
  Change pressure pain threshold in 6 muscles
Algometer Assessment | 3 months of each treatment
  change pressure pain threshold in 6 muscles
Algometer Assessment | 4 months
  change pressure pain threshold in 6 muscles

OTHER OUTCOMES:
Neuropsychological tests | Before each treatment
  Frontal assessment battery
Neuropsychological tests | 3 months of each treatment
  Frontal assessment battery
Neuropsychological tests | 4 months
  Frontal assessment battery
Neuropsychological tests | Before each treatment
  Trail Making Test

CONTACTS AND LOCATIONS:
Locations (1):
- Manuela Deodato, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: Undecided